CLINICAL TRIAL: NCT00346333
Title: Randomized Clinical Trial for Retinitis Pigmentosa
Brief Title: Clinical Trial of Lutein for Patients With Retinitis Pigmentosa Receiving Vitamin A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEI-126
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Results first posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2013-12

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa, Inherited Retinal Degeneration
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Lutein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lutein plus 15,000 IU/d Vitamin A (Experimental): Daily intake of 12mg of Lutein plus 15,000 IU/d of Vitamin A palmitate
  Interventions: Drug: Lutein
- Control plus 15,000 IU/d Vitamin A (Placebo Comparator): Daily intake of cornstarch control plus 15,000 IU/d Vitamin A palmitate
  Interventions: Dietary Supplement: Cornstarch control

INTERVENTIONS:
Drug: Lutein — 12mg/d
  Arms: Lutein plus 15,000 IU/d Vitamin A
Dietary Supplement: Cornstarch control — Daily intake of cornstarch control plus 15,000 IU/d Vitamin A palmitate
  Arms: Control plus 15,000 IU/d Vitamin A

SUMMARY:
The purpose of this trial is to determine whether lutein in addition to vitamin A will slow the course of retinitis pigmentosa.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a group of inherited retinal degenerations with a worldwide prevalence of approximately 1 in 4,000. Patients typically report night blindness and difficulty with mid-peripheral visual field in adolescence. As the condition progresses, they lose far peripheral visual field. Most patients have reductions in central vision by 60 years if left untreated. Vitamin A palmitate, 15,000 International Units (IU)/d and an omega-3 rich diet have been shown to slow the progression of this condition among adults with the typical forms.(see Archives of Ophthalmology,111:761-772,1993 ; Archives of Ophthalmology 122: 1306-1314, 2004; Archives of Ophthalmology 130(6):701-711,2013).

The present study was a randomized, controlled, double-masked trial with a planned duration of 5 years.Two hundred and forty adults with the typical forms of RP were assigned to either lutein 12mg/d or a control group. Patients in both groups received 15,000 IU/day of vitamin A palmitate in addition to the supplement under study. Participants agreed not to know the contents of the supplement or their group assignment until the end of the trial. The main outcome measurement was the total point score for the 30-2 program of the Humphrey Field analyzer (HFA). In addition,the total point score for the 60-4 program ,the total point score of the 30-2 and 60-4 programs combined, computer-averaged 30-Hz cone Electroretinogram (ERG) amplitude and Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity were measured annually as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

Ocular Criteria

* RP, typical forms(i.e. elevated final dark adaptation threshold,retinal arteriolar narrowing,and reduced and delayed full-field ERGs).
* Best-corrected visual acuity 20/100 or better
* HFA program 30-2 total point score >= 250 decibels(dB)to a size V white test light
* No confounding ocular disease such as glaucoma,uveitis,diabetic retinopathy,posterior subcapsular cataract more than 11% of total lens area (ie equivalent to P3 on Lens Opacity Classification System III)and pupil diameter after dilation less than 6 mm.

Dietary Criteria

* Fruit and vegetable intake < 10 servings/d
* Spinach or kale intake < 1 serving/d, i.e. <1/2 cup of cooked spinach or kale per day
* Dietary lutein intake <=5.4 mg/d as estimated from food frequency questionnaire
* No intake of cod liver oil or omega-3 capsules
* Dietary preformed vitamin A intake <= 10,000 IU/d
* Supplement intake <= 5,000 IU/d of Vitamin A and <= 30 IU/d of Vitamin E
* Consumption <= 3 alcoholic beverages/d

Medical and other criteria

* Age 18-60 y
* Body mass index < 40 and weight >= 5th percentile for age,gender,and height
* Serum retinol level <= 100 micrograms/deciliter and serum retinyl ester level <= 380 nanomoles/Liter
* Serum cholesterol < 300 micrograms/deciliter and serum triglyceride level <400 micrograms/deciliter
* No clinically significant abnormality on blood cell count, glucose level, blood urea nitrogen level, serum lipid panel results or serum liver function profile.
* Not pregnant or planning to become pregnant
* Not smoking currently
* Agreed not to know tablet content or course of condition until the end of the trial.
* No other disease which might affect absorption or metabolism of lutein or vitamin A.
* Only one patient per family was accepted into the study.

Exclusion Criteria:

* Women who are pregnant or planning to become pregnant (Vitamin A supplements can increase the risk of birth defects.)
* Current participation in another clinical trial for RP
* Patients with atypical forms such as paravenous RP, pericentral RP, sector RP,unilateral RP,Refsum disease, Bardet-Biedl syndrome, retinitis punctata albescens and cone-rod dystrophy were excluded as were patients with RP and profound congenital deafness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2003-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliot L Berson, MD, Study Chair — Harvard Medical School (HMS and HSDM)
Locations (1):
- Berman Gund Laboratory for the Study of Retinal Degenerations, Harvard Medical School ,Massachusetts Eye & Ear Infirmary, Boston, Massachusetts, United States

REFERENCES:
- [Result] Berson EL, Rosner B, Sandberg MA, Weigel-DiFranco C, Brockhurst RJ, Hayes KC, Johnson EJ, Anderson EJ, Johnson CA, Gaudio AR, Willett WC, Schaefer EJ. Clinical trial of lutein in patients with retinitis pigmentosa receiving vitamin A. Arch Ophthalmol. 2010 Apr;128(4):403-11. doi: 10.1001/archophthalmol.2010.32. PMID 20385935
- [Derived] Comander J, Weigel DiFranco C, Sanderson K, Place E, Maher M, Zampaglione E, Zhao Y, Huckfeldt RM, Bujakowska KM, Pierce E. Natural history of retinitis pigmentosa based on genotype, vitamin A/E supplementation, and an electroretinogram biomarker. JCI Insight. 2023 Aug 8;8(15):e167546. doi: 10.1172/jci.insight.167546. PMID 37261916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We performed screening examinations in the Berman-Gund Laboratory at the Massachusetts Eye & Ear Infirmary, Boston Massachusetts from July 15, 2003 to October 28, 2004.
Pre-assignment Details: We screened patients for eligibility according to ocular, dietary, and medical criteria & performed a baseline examination on eligible patients within 8 weeks. At the baseline visit patients were randomized to 1 of 2 groups taking into account genetic type and initial serum lutein level (<= 6.4 micrograms/deciliter (mg/dL) or > 6.4 mg/dL).
Groups:
- Control Plus Vitamin A: cornstarch control plus 15,000 IU Vitamin A palmitate daily
- Lutein Plus Vitamin A: 12mg Lutein plus 15,000 IU Vitamin A palmitate daily
Period: Overall Study
Arm/Group | Control Plus Vitamin A | Lutein Plus Vitamin A
Started | 121 | 119
Completed | 116 | 111
Not Completed | 5 | 8
Not completed — Death | 1 | 0
Not completed — unwilling or unable to continue | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Control Plus Vitamin A: cornstarch control plus 15,000IU Vitamin A palmitate daily
- Lutein Plus Vitamin A: 12mg Lutein plus 15,000IU Vitamin A palmitate daily
- Total: Total of all reporting groups
Arm/Group | Control Plus Vitamin A | Lutein Plus Vitamin A | Total
Number analyzed (Participants) | 121 | 119 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 121 | 119 | 240
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (1.0) | 40 (1.0) | 39 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 58 | 109
  Male | 70 | 61 | 131
Age of participants by 10-year age groups [Number; unit: Participants]
  18-29 years of age | 34 | 25 | 59
  30-39 years of age | 26 | 35 | 61
  40-49 years of age | 41 | 36 | 77
  50-60 years of age | 20 | 23 | 43
Genetic type [Number; unit: participants]
  Dominant | 30 | 28 | 58
  Recessive | 20 | 19 | 39
  X-Linked | 8 | 7 | 15
  Isolate | 58 | 60 | 118
  Undetermined | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Central Visual Field (vf) Change Assessed Using the 30-2 Program of the Humphrey Field Analyzer (HFA).
Description: Sum of visual field sensitivity readings in decibel(dB) to a size V target out to the 30 degree meridian in each direction of the visual field. The value presented represents annual change in dB over 4 years.
Time Frame: assessed at each of 4 annual visits after baseline
Population: Intention to treat analysis;sample of 215 patients with all 4 years of followup and reliable, non missing data at all 4 years was analyzed. Eyes with an initial 30-2 total point score >= 250 dB were included.The eye was the unit of analysis. Each patient contributed 2,1, or 0 eyes with non-missing data.
Measure: Mean (Standard Error); unit: annual change in db vf sensitivity
Arm/Group | Control Plus Vitamin A | Lutein Plus Vitamin A
Number analyzed (Participants) | 110 | 105
annual change in db vf sensitivity | -51.5 (3.2) | -49.6 (3.3)
Statistical Analysis 1: Comparison: Control Plus Vitamin A vs Lutein Plus Vitamin A; Primary Analysis:Proc mixed of the Statistical Analysis System (SAS) was used to compare annual rates of change by treatment group over 4 years. Power Calculation:240 patients were estimated to be needed to provide sufficient power (i.e. alpha=0.05;beta=0.10)to observe a statistically significant difference between mean change in the 2 groups on the HFA 30-2 total point score over a 4-year interval; Test type: Superiority or Other; p = 0.66, Longitudinal regression analysis — A priori threshold for statistical significance= 0.05. Annual assessments of data by data monitoring board were done with p-values adjusted using the O'Brien-Fleming rule for intermediate looks
Statistical Analysis 2: Comparison: Control Plus Vitamin A vs Lutein Plus Vitamin A; Secondary Analysis: As change distribution was non-normal, slope for each eye was calculated with least squares regression and converted to ranks. The Clustered Wilcoxon test was used to compare slope distributions between groups accounting for correlation between slopes for eyes within individuals; Test type: Superiority or Other; p = 0.52, Clustered Wilcoxon — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Mid-peripheral Field Change Assessed With the 60-4 Program of the Humphrey Field Analyzer.
Description: Sum of visual field sensitivity readings in dB to a size V target from the 30 degree meridian to the 60 degree meridian in each direction of the visual field. The value presented represents annual change in dB over 4 years.
Time Frame: assessed at each of 4 annual visits after baseline
Population: This was an intention to treat analysis;lower sample sizes for this endpoint reflect instances where test results were not available for this outcome variable.The ability to perform this test was not a criterion for study entry.Eyes with an initial score ≥ 10 were included. Values were set to zero for all visits after an initial value of zero.
Measure: Mean (Standard Error); unit: annual change in dB vf sensitivity
Arm/Group | Control Plus Vitamin A | Lutein Plus Vitamin A
Number analyzed (Participants) | 82 | 81
annual change in dB vf sensitivity | -34.1 (3.0) | -26.6 (3.1)
Statistical Analysis 1: Comparison: Control Plus Vitamin A vs Lutein Plus Vitamin A; Primary Analysis: Proc Mixed of SAS was used to compare annual rates of change by treatment group over four years.The unit of analysis was the eye. Each patient contributed 2, 1, or 0 eyes with non-missing data; Test type: Superiority or Other; p = 0.05, Longitudinal regression analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Control Plus Vitamin A vs Lutein Plus Vitamin A; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.03, Clustered Wilcoxon — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Total Field Change Assessed by the Combined 30-2 and 60-4 Programs of the Humphrey Field Analyzer.
Description: Sum of visual field sensitivity readings in dB to a size V target obtained with the 30-2 and 60-4 programs of the Humphrey Field Analyzer combined for those patients on whom both measures were available.
Time Frame: assessed at each of 4 annual visits after baseline
Population: This was an intention to treat analysis. A total field was calculated for each eye using the 30-2 and 60-4 conditions after applying the eligibility criteria for each component. Total field for a given eye was not calculated if either was missing. The unit of analysis was the eye.Each patient contributed 2, 1, or 0 eyes with non-missing data.
Measure: Mean (Standard Error); unit: annual change in dB vf sensitivity
Arm/Group | Lutein Plus Vitamin A | Control Plus Vitamin A
Number analyzed (Participants) | 79 | 78
annual change in dB vf sensitivity | -83.1 (6.2) | -92.9 (5.7)
Statistical Analysis 1: Comparison: Lutein Plus Vitamin A vs Control Plus Vitamin A; Primary analysis:Proc Mixed of SAS was used to compare annual rates of change by treatment group over four years.The unit of analysis was the eye.Each patient contributed 2,1,or 0 eyes with non-missing data; Test type: Superiority or Other; p = 0.24, Longitudinal regression analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Lutein Plus Vitamin A vs Control Plus Vitamin A; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.20, Clustered Wilcoxon — Apriori threshold for statistical significance= 0.05. Annual assessments of data by data monitoring board were done with p-values adjusted using the O'Brien-Fleming rule for intermediate looks

4. Secondary Outcome: Annual Change in 30 Hertz(Hz)Electroretinogram(ERG )Amplitude in Natural Log (ln) Microvolts/yr Over a 4 Year Period.
Description: Computer averaged 30 Hz ERG amplitudes in microvolts for those with initial amplitudes of >= 0.68 microvolts. Presented on the ln scale.
Time Frame: assessed at each of 4 annual visits after baseline
Population: This was an intention to treat analysis;analyses of 30 Hz ERG data included those who had an initial amplitude of 0.68 microvolts or greater in at least 1 eye and data were censored when values declined to less than 0.34 microvolts. The unit of analysis was the eye.Each patient contributed 2,1,or 0 eyes with non-missing data.
Measure: Mean (Standard Error); unit: ln (microvolts)/year
Arm/Group | Control Plus Vitamin A | Lutein Plus Vitamin A
Number analyzed (Participants) | 77 | 79
ln (microvolts)/year | -0.08 (0.12) | -0.09 (0.01)
Statistical Analysis 1: Comparison: Control Plus Vitamin A vs Lutein Plus Vitamin A; Proc MIXED of SAS was used to compare annual rates of change over four years between the treatment groups; Test type: Superiority or Other; p = 0.59, Longitudinal regression analysis — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity
Description: Annual change in number of letters read.
Time Frame: assessed at each of 4 annual visits after baseline
Population: This was an intention to treat analysis and included all reliable, non-missing values. The unit of analysis was the eye.Each patient contributed 2,1, or 0 eyes with non-missing data.
Measure: Mean (Standard Error); unit: Change in letters read per year
Arm/Group | Control Plus Vitamin A | Lutein Plus Vitamin A
Number analyzed (Participants) | 111 | 110
Change in letters read per year | -0.49 (0.12) | -0.53 (0.12)
Statistical Analysis 1: Comparison: Control Plus Vitamin A vs Lutein Plus Vitamin A; Proc MIXED of SAS was used to compare annual rates of change over 4 years between the 2 groups; Test type: Superiority or Other; p = 0.80, Longitudinal regression analysis — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the entire study period. This monitoring included questionnaires at annual visits and over the telephone at 3 month intervals, blood tests at annual visits,and evaluations by the consulting internist if needed.
Groups:
- Control Plus Vitamin A: Daily intake of cornstarch control plus 15,000IU Vitamin A palmitate
- Lutein Plus Vitamin A: 12mg Lutein plus 15,000IU Vitamin A daily.
Arm/Group | Control Plus Vitamin A | Lutein Plus Vitamin A
Serious Adverse Events (participants affected / at risk) | 1/121 | 1/119
Other Adverse Events (participants affected / at risk) | 0/121 | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Plus Vitamin A (N=121) | Lutein Plus Vitamin A (N=119)
Death (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Elevated liver enzymes (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No